CLINICAL TRIAL: NCT01228461
Title: Risk of Fatigue in Adolescent and Young Adult Hodgkin Lymphoma Patients
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 091550
Record Dates: First submitted 2010-10-22; First posted 2010-10-26 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Fatigue; Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma Survivors; Adolescent and Young Adults
MeSH Terms: conditions — Fatigue; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples for IL-1ra and CRP
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AYA with Fatigue and Hodgkin Lymphoma

SUMMARY:
Fatigue is one of the most prevalent symptoms endorsed by cancer survivors, particularly those treated for breast cancer or Hodgkin lymphoma. Despite the tremendous implications such work has for effective interventions, little is known about the underlying pathophysiology of fatigue, association with medical co-morbidities and factors that may help predict those to be at highest risk.

The proposed research will utilize Vanderbilt-Ingram Cancer Center REACH for Survivorship Program together with the investigators Hematologic Malignancies Program. In adolescent and young adults (AYA), ages 18 - 39 the investigators will address the following:

Primary Aims Aim 1: Assess the prevalence and severity of fatigue and its impact on functional outcomes Aim 2: Determine host, disease and treatment-related risk factors for fatigue

Secondary Aims Aim 1: Evaluate the association between levels of proinflammatory cytokine activity and fatigue Aim 2: Evaluate the association between fatigue and self reported fatigue in AYA Hodgkin lymphoma (HL) survivors.

Hypotheses:

1. Fatigue is more prevalent and severe among AYA HL patients and survivors, compared to general population and will be associated with impaired functional outcome.
2. Risk factors for fatigue include higher disease stage, B symptoms and elevated erythrocyte sedimentation rate at diagnosis, dose density of chemotherapy and higher doses and more expanded fields of radiotherapy.
3. Risk of fatigue is associated with long-term cardiopulmonary and endocrine complications.
4. Levels of specified proinflammatory cytokines are associated with increased fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Currently 18 years of age or older
* Alive without evidence of recurrent disease
* Must be off therapy (not on active treatment for HL or other malignancies)
* Must not be on any form of chemotherapy (oral or intravenous [IV])
* Provide informed consent
* Can read and understand English
* Treated with risk-adapted therapy which may include radiotherapy doses < 30 Gy

Exclusion Criteria:

* Evidence of a subsequent malignancy following lymphoma treatment

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adult survivors of Hodgkin Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Prevalence and severity of fatigue and its impact on functional outcomes | 1 year

SECONDARY OUTCOMES:
Evaluate the association between levels of proinflammatory cytokine activity and fatigue | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States